CLINICAL TRIAL: NCT03552276
Title: A Long-Term Extension Study to Demonstrate Safety of Tildrakizumab in Subjects With Psoriatic Arthritis Who Have Previously Completed Study With Tildrakizumab.
Brief Title: Long-Term Extension Trial of Tildrakizumab to Prove Its Safety in Subjects With Psoriatic Arthritis Who Have Previously Completed Study With Tildrakizumab.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CLR_18_07
Record Dates: First submitted 2018-05-04; First posted 2018-06-11 (Actual); Results first posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-10

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — tildrakizumab

STUDY DESIGN:
Masking Description: Subjects will be not be randomized and will enter the long-term extension study with one fixed dose regimen of tildrakizumab, low dose regimen at Week 52 of the parent study.
  Study was double blind until Databaselock of parent study happened to maintain blinding Subjects continue to assigned treatment from parent study up to week 52 in the Long term extension and there after all subjects began migrating to receive low dose injection Q12 weeks in an open-label fashion for up to an additional 4 years..
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- SUNPG18_07 q4 weeks, high dose (Experimental): Tildrakizumab 200 mg q4 Weeks
  Interventions: Drug: SUNPG18_07 I (Tildrakizumab 200 mg)
- SUNPG18_07 q12 weeks, high dose (Experimental): Tildrakizumab 200 mg q12 Weeks
  Interventions: Drug: SUNPG18_07 I (Tildrakizumab 200 mg)
- SUNPG18_07 q12 weeks, low dose (Experimental): Tildrakizumab 100 mg q12 Weeks
  Interventions: Drug: SUNPG18_07 II (Tildrakizumab 100 mg)
- SUNPG18_07 q4 Weeks, High Dose to SUNPG18_07 q12 Weeks, Low Dose (Experimental): Tildrakizumab 200 mg q4 weeks switched to tildrakizumab 100 mg q12 weeks
  Interventions: Drug: SUNPG18_07 I (Tildrakizumab 200 mg); Drug: SUNPG18_07 II (Tildrakizumab 100 mg)
- SUNPG18_07 q12 Weeks, High Dose to SUNPG18_07 q12 Weeks, Low Dose (Experimental): Tildrakizumab 200 mg q12 weeks switched to tildrakizumab 100 mg q12 weeks
  Interventions: Drug: SUNPG18_07 I (Tildrakizumab 200 mg); Drug: SUNPG18_07 II (Tildrakizumab 100 mg)

INTERVENTIONS:
Drug: SUNPG18_07 I (Tildrakizumab 200 mg) — injection
  Arms: SUNPG18_07 q12 Weeks, High Dose to SUNPG18_07 q12 Weeks, Low Dose; SUNPG18_07 q12 weeks, high dose; SUNPG18_07 q4 Weeks, High Dose to SUNPG18_07 q12 Weeks, Low Dose; SUNPG18_07 q4 weeks, high dose
Drug: SUNPG18_07 II (Tildrakizumab 100 mg) — injection
  Arms: SUNPG18_07 q12 Weeks, High Dose to SUNPG18_07 q12 Weeks, Low Dose; SUNPG18_07 q12 weeks, low dose; SUNPG18_07 q4 Weeks, High Dose to SUNPG18_07 q12 Weeks, Low Dose

SUMMARY:
A long term study to demonstrate the safety of Tildrakizumab in Subjects with Psoriatic Arthritis who Have Previously Completed Study with Tildrakizumab

DETAILED DESCRIPTION:
Subjects have rolled over from parent study, i.e., CLR_16_23, into the long-term extension study CLR_18_07.

The study has been open label post 1 year completion.

ELIGIBILITY:
Inclusion Criteria:

Subjects may be included in the study if they meet all of the following criteria:

1. Subject has provided written informed consent for this long-term extension study.
2. Subjects with PsA who met the inclusion criteria of the parent study and completed the parent study treatment period (e.g., up to Week 48 for the parent Phase 2 study, with return for the EoT assessment at Week 52).
3. No concomitant use of both leflunomide and methotrexate,
4. No history of active tuberculosis (TB) or symptoms of TB.

Exclusion Criteria:

Subjects should be excluded from the study if they meet any of the following criteria:

1. New onset during the parent study of arthritic conditions other than the subject's original condition.
2. Female subjects of childbearing potential who do not agree to abstain from heterosexual activity or practice a dual method of contraception, for example, a combination of the following: (1) oral contraceptive, depo-progesterone, or intrauterine device; and (2) a barrier method (condom or diaphragm). Male subjects with female partners of childbearing potential who are not using birth control as described above must use a barrier method of contraception (e.g., condom) if not surgically sterile (i.e., vasectomy). Contraceptive methods must be practiced upon entering the study and through 16 weeks after the last dose of IMP. If a subject discontinues prematurely, the contraceptive method must be practiced for 16 weeks following final administration of IMP.
3. Female is pregnant or breastfeeding, or planning to become pregnant or initiate breastfeeding while enrolled in the study or up to 16 weeks after the last dose of IMP.
4. Subject has previously been enrolled in this long-term extension study.
5. Any condition that in the opinion of the Investigator represents an obstacle for study conduct and/or represents a potential unacceptable risk for the subject.
6. Subject has any concurrent medical condition or uncontrolled, clinically significant systemic disease (e.g., renal failure, heart failure, hypertension, liver disease, diabetes, or anemia) that, in the opinion of the Investigator, could cause continued treatment to be detrimental to the subject.
7. Subject has a known history of infection with hepatitis B, hepatitis C, or human immunodeficiency virus during the parent study.
8. Subjects with a history of alcohol or drug abuse during the parent study.
9. Subject has a need for use of a live vaccine within 10 weeks of final anticipated dose of IMP for the long-term extension study.
10. Concomitant use of prohibited medications or use of commercially available or investigational biologic therapies (other than tildrakizumab) for PsO and/or PsA
11. Subjects who have been placed in an institution on official or judicial orders.
12. Subjects who are related to or dependent on the Investigator, Sponsor, or study site such that a conflict of interest may arise.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2023-09-18 (Actual); Study Completion 2023-09-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (66):
- United States (13):
  - Site 25, Glendale, Arizona
  - Site 16, Phoenix, Arizona
  - Site 14, Denver, Colorado
  - Site 27, Wichita, Kansas
  - Site 23, Lexington, Kentucky
  - Site 20, Monroe, Louisiana
  - Site 26, Lebanon, New Hampshire
  - Site 24, Salisbury, North Carolina
  - Site 19, Cincinnati, Ohio
  - Site 17, Middleburg Heights, Ohio
  - Site 18, Memphis, Tennessee
  - Site 21, Seattle, Washington
  - Site 22, Spokane, Washington
- Argentina (3):
  - Site 02, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Site 01, Mar del Plata, Buenos Aires
  - Site 03, San Fernando, Buenos Aires
- Hungary (3):
  - Site 32, Budapest
  - Site 34, Budapest
  - Site 33, Kistarcsa
- Mexico (10):
  - Site 09, Mexico City, Mexico City
  - Site 05, Mexico City, Mexico City
  - Site 06, Monterrey, Nuevo León
  - Site 13, San Luis Potosí City, San Luis Potosí
  - Site 04, San Luis Potosí City, San Luis Potosí
  - Site 07, Culiacán, Sinaloa
  - Site 12, Mérida, Yucatán
  - Site 11, Chihuahua City
  - Site 08, Cuautitlán Izcalli
  - Site 10, Durango
- Poland (14):
  - Site 45, Krakow, Lesser Poland Voivodeship
  - Site 38, Bialystok
  - Site 47, Bytom
  - Site 36, Elblag
  - Site 39, Katowice
  - Site 40, Katowice
  - Site 46, Krakow
  - Site 43, Lodz
  - Site 48, Nowa Sól
  - Site 42, Poznan
  - Site 53, Sochaczew
  - Site 50, Warsaw
  - Site 52, Warsaw
  - Site 51, Wroclaw
- Russia (9):
  - Site 61, Kemerovo, Kemerovo Oblast
  - Site 58, Novosibirsk, Novosibirsk Oblast
  - Site 54, Tomsk, Tomsk Oblast
  - Site 56, Izhevsk
  - Site 60, Moscow
  - Site 57, Saint Petersburg
  - Site 62, Smolensk
  - Site 55, Yaroslavl
  - Site 59, Yaroslavl
- Spain (6):
  - Site 67, Santiago de Compostela, La Coruna
  - Site 65, Málaga, Malaga
  - Site 68, Bilbao, Vizcaya
  - Site 66, Barcelona
  - Site 64, Barcelona
  - Site 71, Seville
- Ukraine (8):
  - Site 75, Kharkiv
  - Site 73, Kiev
  - Site 74, Kyiv
  - Site 76, Kyiv
  - Site 72, Kyiv
  - Site 77, Odesa
  - Site 79, Vinnytsia
  - Site 78, Zaporizhzhia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a long-term extension (LTE) study in subjects with Psoriatic arthritis who had completed the treatment with tildra in the parent study,CLR_16_23(NCT02980692). In LTE, there was no randomization and subjects continued to receive the treatment assigned during the parent study into the LTE upto Wk 52 to maintain blind of the parent study. Post the DBL of CLR 16-23, the blind was no longer needed, all subjects who had entered the LTE study received open label dose of tildra 100 mg q12 wks.
Groups:
- Tildrakizumab 200 mg q4 Weeks; Tildrakizumab 200 mg q12 Weeks: The subjects in this group entered the LTE study from the parent study, however, they discontinued from the study and were not switched to the open label tildrakizumab 100 mg q12 weeks dose.
- Tildrakizumab 100 mg q12 Weeks: These subjects continued to receive same dose of tildrakizumab 100 mg q12 weeks in the LTE study as in the parent study. However, in the LTE study, post DBL of the parent study, the dose was open label
- Tildrakizumab 200 mg q4 Weeks Switched to Tildrakizumab 100 mg q12 Weeks: This group represents subjects who switched from tildrakizumab 200 mg q4 weeks dose to open label tildrakizumab 100 mg q12 weeks dose in the LTE study, post DBL of the parent study.
- Tildrakizumab 200 mg q12 Weeks Switched to Tildrakizumab 100 mg q12 Weeks: This group represents subjects who switched from tildrakizumab 200 mg q12 weeks dose to open label tildrakizumab 100 mg q12 weeks dose in the LTE study, post DBL of the parent study
Period: Overall Study
Arm/Group | Tildrakizumab 200 mg q4 Weeks | Tildrakizumab 200 mg q12 Weeks | Tildrakizumab 100 mg q12 Weeks | Tildrakizumab 200 mg q4 Weeks Switched to Tildrakizumab 100 mg q12 Weeks | Tildrakizumab 200 mg q12 Weeks Switched to Tildrakizumab 100 mg q12 Weeks
Started | 5 | 22 | 49 | 54 | 151
Completed | 0 | 0 | 33 | 46 | 126
Not Completed | 5 | 22 | 16 | 8 | 25

BASELINE CHARACTERISTICS:
Groups:
- Tildrakizumab q4 Weeks, 200 mg; Tildrakizumab 200 mg q12 Weeks: The subjects in this group entered the LTE study from the parent study, however, they discontinued from the study and were not switched to the open label tildrakizumab 100 mg q12 weeks dose.
- Total: Total of all reporting groups
Arm/Group | Tildrakizumab q4 Weeks, 200 mg | Tildrakizumab 200 mg q12 Weeks | Tildrakizumab 100 mg q12 Weeks | Tildrakizumab 200 mg q4 Weeks Switched to Tildrakizumab 100 mg q12 Weeks | Tildrakizumab 200 mg q12 Weeks Switched to Tildrakizumab 100 mg q12 Weeks | Total
Number analyzed (Participants) | 5 | 22 | 49 | 54 | 151 | 281
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.0 (11.96) | 53.8 (14.80) | 50.6 (11.35) | 49.9 (13.47) | 48.3 (11.93) | 49.7 (12.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 13 | 28 | 33 | 77 | 152
  Male | 4 | 9 | 21 | 21 | 74 | 129
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 6 | 6 | 22 | 39
  Not Hispanic or Latino | 3 | 19 | 43 | 48 | 129 | 242
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 0 | 2 | 4
  White | 5 | 21 | 48 | 53 | 147 | 274
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Please refer to Adverse event section for more information
Time Frame: upto week 208
Measure: Count of Participants; unit: Participants
Arm/Group | Tildrakizumab 200 mg q4 Weeks | Tildrakizumab 200 mg q12 Weeks | Tildrakizumab 100 mg q12 Weeks | Tildrakizumab 200 mg q4 Weeks Switched to Tildrakizumab 100 mg q12 Weeks | Tildrakizumab 200 mg q12 Weeks Switched to Tildrakizumab 100 mg q12 Weeks
Number analyzed (Participants) | 5 | 22 | 49 | 54 | 151
Participants | 5 | 14 | 36 | 44 | 125

ADVERSE EVENTS:
Time Frame: Week 208
Description: The subjects rolled over to the LTE study from the parent study (CLR-16-23) continued to receive the dose as per the parent study upto Week 52 to ensure that blinding of the parent study is maintained. Thereafter, once the data base lock (DBL) of the parent study occurred and the blinding was no longer needed subjects received open label tildrakizumab 100 mg q12 weeks.
Groups:
- Tildrakizumab 200 mg, q4 Weeks: The subjects in this group entered the LTE, however, they discontinued from the study and were not switched to the open label tildrakizumab 100 mg q12 weeks dose.
- Tildrakizumab 200 mg, q12 Weeks: The subjects in this group entered the LTE study, however, they discontinued from the study and were not switched to the open label tildrakizumab 100 mg q12 weeks dose.
- Tildrakizumab 100 mg q12 Weeks: These subjects continued to receive same dose of tildrakizumab 100 mg q12 weeks in the LTE study as in the parent study. However, in the LTE, post DBL of the parent study, the dose was open label.
- Tildrakizumab 200 mg q4 Weeks, to Tildrakizumab 100 mg q12 Weeks; Tildrakizumab 200 mg q12 Weeks, to Tildrakizumab 100 mg q12 Weeks: This group represents subjects who switched from tildrakizumab 200 mg q4 weeks to open label tildrakizumab 100 mg q12 weeks dose in the LTE study, post DBL of the parent study.
Arm/Group | Tildrakizumab 200 mg, q4 Weeks | Tildrakizumab 200 mg, q12 Weeks | Tildrakizumab 100 mg q12 Weeks | Tildrakizumab 200 mg q4 Weeks, to Tildrakizumab 100 mg q12 Weeks | Tildrakizumab 200 mg q12 Weeks, to Tildrakizumab 100 mg q12 Weeks
All-Cause Mortality (participants affected / at risk) | 0/5 | 1/22 | 0/49 | 0/54 | 1/151
Serious Adverse Events (participants affected / at risk) | 3/5 | 2/22 | 7/49 | 3/54 | 25/151
Other Adverse Events (participants affected / at risk) | 5/5 | 14/22 | 36/49 | 44/54 | 125/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tildrakizumab 200 mg, q4 Weeks (N=5) | Tildrakizumab 200 mg, q12 Weeks (N=22) | Tildrakizumab 100 mg q12 Weeks (N=49) | Tildrakizumab 200 mg q4 Weeks, to Tildrakizumab 100 mg q12 Weeks (N=54) | Tildrakizumab 200 mg q12 Weeks, to Tildrakizumab 100 mg q12 Weeks (N=151)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 2
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Abdominal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Gallbladder empyema (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Intestinal sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Biopsy kidney (Investigations) | 0 | 0 | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Retinal migraine (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
End stage renal disease (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Hydrocele female (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Gastric bypass (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
Aortic dissection (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Arteriosclerosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 2
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 2
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tildrakizumab 200 mg, q4 Weeks (N=5) | Tildrakizumab 200 mg, q12 Weeks (N=22) | Tildrakizumab 100 mg q12 Weeks (N=49) | Tildrakizumab 200 mg q4 Weeks, to Tildrakizumab 100 mg q12 Weeks (N=54) | Tildrakizumab 200 mg q12 Weeks, to Tildrakizumab 100 mg q12 Weeks (N=151)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 3
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 2
Neutrophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 2 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Diastolic dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 2
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Pericardial cyst (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Tricuspid valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Accessory spleen (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1
Gilbert's syndrome (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1
Hydrocele (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 1
Autoimmune thyroiditis (Endocrine disorders) | 0 | 0 | 1 | 0 | 0
Goitre (Endocrine disorders) | 0 | 0 | 1 | 1 | 0
Hypothyroidic goitre (Endocrine disorders) | 0 | 0 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1 | 0 | 1
Thyroid mass (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Astigmatism (Eye disorders) | 0 | 0 | 0 | 0 | 1
Blepharitis (Eye disorders) | 0 | 0 | 0 | 0 | 1
Blindness transient (Eye disorders) | 0 | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 1 | 0 | 2
Cataract nuclear (Eye disorders) | 0 | 0 | 0 | 1 | 0
Diabetic retinopathy (Eye disorders) | 0 | 0 | 1 | 0 | 0
Keratitis (Eye disorders) | 0 | 0 | 0 | 0 | 1
Myopia (Eye disorders) | 0 | 0 | 0 | 0 | 1
Retinal vascular disorder (Eye disorders) | 0 | 0 | 0 | 1 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 4 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Abdominal rigidity (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Barrett's oesophagus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Chronic gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1
Coeliac artery stenosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 0 | 3 | 1 | 1
Diaphragmatic hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 4 | 3 | 4 | 6
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 2
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Gingival swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Intestinal metaplasia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 2 | 2 | 0 | 6
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Rectal polyp (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Retained deciduous tooth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 3
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 2
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 2
Chills (General disorders) | 0 | 0 | 0 | 1 | 1
Drug intolerance (General disorders) | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 1 | 0 | 4
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 2 | 0 | 0
Injection site erythema (General disorders) | 0 | 0 | 1 | 2 | 1
Injection site pain (General disorders) | 0 | 0 | 1 | 1 | 2
Injection site pruritus (General disorders) | 0 | 0 | 1 | 1 | 0
Injection site rash (General disorders) | 0 | 0 | 0 | 0 | 1
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 1
Injury associated with device (General disorders) | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 2
Pyrexia (General disorders) | 0 | 0 | 3 | 4 | 4
Vaccination site pain (General disorders) | 0 | 0 | 1 | 0 | 0
Xerosis (General disorders) | 0 | 1 | 0 | 0 | 0
Biliary dyskinesia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Diabetic hepatopathy (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Gallbladder polyp (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 2
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 3
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 1 | 0 | 2
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Steatohepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Allergy to arthropod bite (Immune system disorders) | 0 | 0 | 0 | 0 | 3
Allergy to plants (Immune system disorders) | 0 | 0 | 0 | 0 | 1
Abdominal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Adenovirus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Bacteriuria (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Bartholin's abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Breast abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 2 | 1 | 2 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 3 | 11 | 25
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 3
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Chronic sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 1 | 0 | 1 | 1
Coronavirus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 3
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Erythema migrans (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Escherichia infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Furuncle (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gallbladder empyema (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 3
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Gastrointestinal bacterial overgrowth (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gingivitis (Infections and infestations) | 0 | 0 | 1 | 0 | 2
Helicobacter gastritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Helicobacter infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 1 | 1 | 4
Intestinal sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Joint abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 7 | 8 | 21
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Periodontitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 2 | 9
Pharyngotonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 4
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pulpitis dental (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Purulent discharge (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 2 | 2
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 3 | 1 | 2
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 1 | 13
Septic shock (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 2 | 0 | 2 | 4
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Suspected COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1 | 2
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Tracheitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Tracheobronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 7 | 9 | 13
Urinary tract infection (Infections and infestations) | 1 | 1 | 2 | 3 | 18
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 2
Viral pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Burns second degree (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 3
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Cuboid syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 3
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Iliotibial band syndrome (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Immunisation reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 4
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 2
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 2
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 3
Nail avulsion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Post vaccination syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Synovial rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Tendon injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 2 | 2 | 3
Apolipoprotein B increased (Investigations) | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 2 | 1 | 3
Bilirubin conjugated increased (Investigations) | 0 | 0 | 1 | 0 | 0
Bilirubin urine present (Investigations) | 0 | 1 | 0 | 0 | 0
Biopsy kidney (Investigations) | 0 | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 1 | 0 | 1
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 2 | 3
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 2 | 1 | 3
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 1 | 1
Blood glucose increased (Investigations) | 0 | 0 | 2 | 0 | 0
Blood pressure increased (Investigations) | 1 | 0 | 3 | 0 | 2
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 1
C-reactive protein increased (Investigations) | 0 | 0 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 1 | 1 | 5
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Haematocrit decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 1 | 0 | 1
Low density lipoprotein increased (Investigations) | 0 | 0 | 0 | 1 | 3
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Monocyte count decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Prostatic specific antigen increased (Investigations) | 0 | 0 | 0 | 2 | 0
Red blood cell count decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 1 | 0 | 0
Urinary casts (Investigations) | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Weight increased (Investigations) | 0 | 1 | 0 | 3 | 7
White blood cell count decreased (Investigations) | 0 | 0 | 1 | 1 | 0
Cholesterosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Copper deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 2 | 2 | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 4
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 1 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 2
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 3
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 4
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Impaired fasting glucose (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Insulin resistance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 1 | 3 | 3
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 6
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 1 | 6
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 2 | 6
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2
Dactylitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Fracture pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Greater trochanteric pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 2
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Jaw cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Joint contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 2 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 2 | 2
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 2
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Periarticular disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 1 | 9
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 2
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Spinal disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 2 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 2
Benign oesophageal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 0
Anosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Bradykinesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 2
Cervicobrachial syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Diabetic neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 3 | 4 | 13
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Lumbar radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Lumbosacral radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Myotonia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Neuritis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Parkinson's disease (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 2 | 0 | 0
Retinal migraine (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 1 | 4
Sensory loss (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Spinal cord haematoma (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Adjustment disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Affective disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 2 | 1 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 3
Insomnia (Psychiatric disorders) | 0 | 2 | 0 | 0 | 1
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Mixed anxiety and depressive disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Stress (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 3
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Cystitis noninfective (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1
End stage renal disease (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Glomerulonephritis chronic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Hypertonic bladder (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0
Nephrosclerosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 3
Renal cyst (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1
Stress urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Urinary tract inflammation (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Abnormal uterine bleeding (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Adenomyosis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Bartholin's cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Hydrocele female (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Menstruation irregular (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Prostatomegaly (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 5
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 2
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0
Gastric bypass (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
Aortic arteriosclerosis (Vascular disorders) | 0 | 0 | 0 | 1 | 2
Aortic dissection (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Arteriosclerosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Bleeding varicose vein (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Blood pressure fluctuation (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 2
Diabetic microangiopathy (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Essential hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 2 | 0 | 2 | 5 | 10
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Lymphostasis (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Peripheral venous disease (Vascular disorders) | 0 | 0 | 0 | 1 | 2
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-07-22): https://cdn.clinicaltrials.gov/large-docs/76/NCT03552276/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-11): https://cdn.clinicaltrials.gov/large-docs/76/NCT03552276/SAP_001.pdf